CLINICAL TRIAL: NCT06991192
Title: ACL Reconstruction Rehabilitation With Exercise and Psychological Support
Acronym: ACLR-REPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A23-019; R21AR082572 (NIH)
Record Dates: First submitted 2025-04-21; First posted 2025-05-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: ACL Reconstruction; Anterior Cruciate Ligament; Rehabilitation; Psychological
MeSH Terms: interventions — Rehabilitation; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rehabilitation (No Intervention): TRIA rehabilitation protocols for ACL reconstruction with bone-patellar tendon-bone autograft or ACL reconstruction with meniscal repair will be used for prescribing exercise. Physical therapists may use adjunctive modalities such as neuromuscular electrical stimulation, blood flow restriction, manual therapy, and cryotherapy at their discretion. Exercise videos prescribed to study participants will be housed in an individual online account per standard clinical procedure (MedBridge, Bellevue, WA).
- Psychological Support (REPS) (Experimental): Study participants in Rehabilitation with Exercise and Psychological Support (REPS) will receive the standard rehabilitation treatment AND psychological support through a combination of PT training and patient training videos.
  Interventions: Behavioral: Rehabilitation with Exercise and Psychological Support (REPS)

INTERVENTIONS:
Behavioral: Rehabilitation with Exercise and Psychological Support (REPS) — Rehabilitation with Exercise and Psychological Support (REPS) is a rehabilitation approach that integrates exercise with psychological support provided by physical therapist and patient training videos.
  Arms: Psychological Support (REPS)

SUMMARY:
The purpose of this study is to examine ACLR Rehabilitation with Exercise and Psychological Support (REPS), comparing two approaches for providing psychological support along with exercise during ACL reconstruction rehabilitation. In one group, physical therapists have received training that may boost emotional support during rehabilitation. In the other group, physical therapists will not have the training. Both groups will get similar exercises and participate in the same testing. Both groups will also watch short videos during rehabilitation that are specific to their group. Participants will not know to which group they are assigned until the end of the study. Participation will attend a total of four study visits over the course of 6 months, including 1 visit before the surgery and 3 visits during follow-up.

DETAILED DESCRIPTION:
The objective of this study is to examine the efficacy of Rehabilitation with Exercise and Psychological Support (REPS), a rehabilitation approach that integrates exercise with psychological support provided by physical therapist and patient training videos. The central hypothesis is that REPS will facilitate better psychological response (Specific Aim 1) and knee function (Specific Aim 2) than Standard Rehabilitation after ACL reconstruction. The feasibility, acceptability, and fidelity of implementing REPS will be explored. This is a pilot randomized controlled trial of 60 patients with ACL reconstruction who receive REPS or Standard Rehabilitation. Study participants in both treatment arms will receive exercise per a standard rehabilitation protocol. Physical therapists providing the REPS intervention will receive didactic training in psychologically informed practice principles and REPS procedures, clinical application practice, and regular feedback from the study team. Study participants in REPS will receive training videos on psychosocial aspects of recovery and mental skills to improve the psychological response. Study visits will occur prior to surgery (baseline), immediately before the first rehabilitation visit post-surgery, 3 months post-surgery, and 6 months post-surgery.

Study Aims Specific Aim 1. To examine the efficacy of REPS on psychological response after ACL reconstruction. Primary Hypothesis: Psychological readiness for sport, measured with the ACL Return to Sport after Injury (ACL-RSI) scale, will be higher in REPS than Standard Rehabilitation at 6 months post-surgery. Secondary Hypothesis: Kinesiophobia, measured with the Tampa Scale for Kinesiophobia (TSK-11) questionnaire, will be lower in REPS than Standard Rehabilitation at 6 months post-surgery.

Specific Aim 2. To examine the efficacy of REPS on knee function after ACL reconstruction. Hypothesis: Self-reported knee function, measured with the International Knee Documentation Committee (IKDC) subjective form, will be higher in REPS than Standard Rehabilitation at 6 months post-surgery.

Exploratory Aim. To assess the feasibility, acceptability, and fidelity of implementing REPS after ACL reconstruction. Research records will be used to assess the feasibility of REPS, and develop surveys for patients and clinicians will be used to assess the acceptability of REPS. In both treatment arms, patients will complete questionnaires that align with anticipated clinical changes in empathy (Consultation and Relational Empathy, CARE) and therapeutic alliance (Working Alliance Inventory-Short Revised, WAI-SR), and documentation templates will be used to record treatments and training for descriptive analysis of fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 21 years at the time of surgery;
* Pre-injury Tegner Activity Rating60 ≥ 5 (5=recreational sports, 10=elite sports);
* Sports participation at least 100 hours/year prior to injury;
* Intent to resume a pre-injury sport that requires cutting, jumping, or pivoting;
* ACL reconstruction performed ≤ 6 months from injury;
* ACL reconstruction performed with bone-patellar tendon-bone autograft or quadriceps tendon autograft; and
* Able to complete rehabilitation at one of the 4 participating TRIA locations.

Exclusion Criteria:

* Previous ACL injury or surgery to either limb;
* Concomitant ligamentous injury > Grade II or requiring surgery; and
* Surgical procedure to articular cartilage requiring non-weight-bearing after surgery.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
ACL Return to Sport after Injury (ACL-RSI) | Pre-surgery (baseline), prior to first post-surgical rehabilitation visit , 3-months post-surgery, 6-months post-surgery
  The ACL Return to Sport after Injury (ACL-RSI) scale has 12-items in the domains of emotions, confidence, and risk appraisal. Scores range from 0 to 100, and higher scores indicate greater psychological readiness for sport. ACL-RSI has acceptable validity and test-retest reliability.
International Knee Documentation Committee (IKDC) Subjective Form | Pre-surgery (baseline), prior to first post-surgical rehabilitation visit , 3-months post-surgery, 6-months post-surgery
  International Knee Documentation Committee (IKDC) subjective form assesses self-reported knee symptoms and function. It is responsive and reliable across knee pathologies, including ACL reconstruction, and has been used as an outcome in federally-funded ACL reconstruction registries and clinical trials. IKDC scores range from 0 to 100 points, and higher scores indicate better knee function.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Pre-surgery (baseline), prior to first post-surgical rehabilitation visit , 3-months post-surgery, 6-months post-surgery
  TSK-11 has 11-items on kinesiophobia, or pain-related fear of movement/re-injury. Scores range from 11 to 44 points, and higher scores indicate greater kinesiophobia. TSK-11 has demonstrated validity for patients with ACL reconstruction.
Clinical Test (Knee pain) | 3-months and 6-months post-surgery
  The Numeric Pain Rating Scale (NPRS) will be used to assess pain at rest and pain with a countermovement jump, if applicable. The scale ranges from 0 (no pain) to 10 (highest imaginable pain).
Clinical Test (Knee range of motion) | 3-months and 6-months post-surgery
  Knee range of motion (flexion and extension) will be assessed bilaterally in a supine position with a goniometer. Interlimb symmetry will be computed as (non-surgical knee motion - surgical knee motion).
Clinical Test (Quadriceps strength) | 3-months and 6-months post-surgery
  Isometric quadriceps strength will be measured bilaterally on an isokinetic dynamometer (CSMi Solutions, Stoughton, MA) with the knee in 60° of flexion. Peak knee extensor torque (N-m) from 3 trials will be recorded. The interlimb symmetry index for isometric quadriceps strength will be computed as [(surgical limb measure/non-surgical limb measure) * 100].
Clinical Test (Countermovement jump) | 6-months post-surgery
  If the study participant meets clinical criteria, a countermovement jump will be performed on a force platform (Hawkin Dynamics, Westbrook, ME). Jump height, bilateral braking impulse index, bilateral propulsion impulse index, modified reaction strength index and landing stiffness will be recorded.
Clinical Test (Single leg hop battery) | 6-months post surgery
  Single leg hop testing will include three hop tests: single hop, triple crossover hop, and lateral timed hop. Subjects will receive verbal instruction and visual demonstration followed by 1 or more practice trials. Subjects will then perform three test trials on each leg, and the best performance (distance or time) will be recorded and expressed as a percentage (involved/uninvolved x 100). This outcome will be calculated as the average limb symmetry index across the three tests with scores ranging from 0 to 100. Higher scores reflect better symmetry and increased function.
Clinical Test (Squat test) | 3-months post-surgery
  Patient will stand on a force plate and perform a squat. Two trials will be collected and two metrics will be reported Left/right average force asymmetry (%) and Left/right peak force asymmetry (%).

OTHER OUTCOMES:
Feasibility: Enrollment Rate | From the date when study enrollment was initiated until the last study participant is enrolled, up to 24 months
  Feasibility of implementing REPS after ACL reconstruction will be measured by calculating the percentage of patients who enrolled in the trial from the number screened for eligibility. This will be reported as a single point estimate with the denominator being the number of patients screened, larger than the sample size used for other outcome measures.
Feasibility: Drop-out Rate | From enrollment to 6-months post-surgery
  Feasibility of of implementing REPS after ACL reconstruction will be measured by calculating the percentage of enrolled patients who withdraw from the study before the end of the intervention period.
Acceptability: REPS Patient Experience | 6-months post-surgery
  Patient reported acceptability of implementing REPS after ACL reconstruction will be assessed from responses to the question "I like learning about how my mind responds to my injury" as part of the 6-month post-surgery REPS patient experience survey. The percentage of REPS intervention patients who report either "Strongly agree" or "Somewhat agree" will be reported. This outcome will only be measured in patient randomized to the REPS study arm.
Fidelity (Receipt): Consultation and Relational Empathy (CARE) | 3-months and 6-months post-surgery
  The Consultation and Relational Empathy (CARE) measure is a 10-item patient-assessed questionnaire that captures empathetic support provided for patients in clinical and general medical settings. Items assess how well the patient felt their doctor listened, was positive and compassionate. CARE scores range from 1 to 50 points, and higher scores indicate higher empathy in the consultation process.
Fidelity (Receipt): Working Alliance Inventory-Short Revised (WAI-SR) | 3-months and 6-months post-surgery
  The Working Alliance Inventory-Short Revised (WAI-SR) measure is a 12-item patient-assessed questionnaire that captures key aspect of the therapeutic alliance. WAI-SR scores range from 15 to 60 points, and higher scores indicate stronger therapeutic alliance.
Fidelity (Delivery): Rehabilitation Dose | From initial rehabilitation visit to 6-months post-surgery
  Delivery of patient training will be measured throughout the post-surgery period via proportion of scheduled visits attended. The average attendance will be summarized from treatment documentation templates in the electronic medical record at 6 months post-surgery and calculated separately for the REPS and comparison arms.

CONTACTS AND LOCATIONS:
Locations (1):
- TRIA, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No